CLINICAL TRIAL: NCT02275000
Title: Randomised Feasibility Study of a Physiotherapy Programme for Patients With Functional Motor Symptoms (FMS).
Brief Title: Feasibility Study of Physiotherapy for Functional Motor Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14/LO/0573
Record Dates: First submitted 2014-10-20; First posted 2014-10-27 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2015-05

CONDITIONS: Conversion Disorder
MeSH Terms: conditions — Conversion Disorder | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): 5 Day physiotherapy programme at the National Hospital for Neurology and Neurosurgery, Queen Square, London UK.
  Interventions: Other: 5 Day Physiotherapy Programme
- Treatment as usual (Active Comparator): Participants are referred to their local neuro-physiotherapy service and if appropriate placed on a waiting list for inpatient rehabilitation.
  Interventions: Other: Physiotherapy

INTERVENTIONS:
Other: 5 Day Physiotherapy Programme — The experimental group will complete a 5 day physiotherapy programme consisting of education, movement retraining and a self management plan.
  Arms: Intervention
Other: Physiotherapy — Treatment as usual physiotherapy. The participant will be referred to their closest NHS outpatient neuro-physiotherapy service.
  Arms: Treatment as usual

SUMMARY:
The aim of this study is to develop and assess the feasibility of a physiotherapy intervention for people with functional motor symptoms (also known as psychogenic neurological symptoms and conversion disorder). Participants will be randomised to receive the intervention or a "treatment as usual" control.

DETAILED DESCRIPTION:
Participants will be recruited from outpatient neurology clinics at Queen Square. Those who consent to take part will complete baseline outcome measures (Time 1) before being randomised to either a Treatment as Usual control group or the Intervention group.

Treatment as Usual group -

1. Participants will be directed to online patient information resources (www.neurosymptoms.org)
2. Participants will be placed on the waiting list to be assessed for the inpatient treatment programme for functional symptoms at The National Hospital for Neurology and Neurosurgery. The waitlist is currently greater than 12 months.
3. A referral is made to local community therapy services (which may include physiotherapy, occupational therapy and psychological therapy). If the participant has had contact from their community therapy services in the previous 12 months, a letter summarising the participant's diagnosis and physiotherapy needs will be sent.
4. Participants will be asked to return at 4 weeks to complete outcome measures for a second time (Time 2)

A referral to community therapy for such patients is usual practice in the UK, although the form in which the community therapy is provided tends to be inconsistent across the UK. In most cases it will entail between 1 and 8 outpatient or domiciliary physiotherapy appointments. Some communities will have access to Occupational Therapy, which may entail supported practice and advice to increase independence with functional tasks and the provision of equipment. The provision of community therapy to participants will be monitored through the CSRI.

Intervention Group -

For participants allocated to the intervention group, a 5 day admission on the Day Hospital at the National Hospital for Neurology and Neurosurgery is arranged. The physiotherapy intervention will take place in the physiotherapy department. Participants will be admitted individually (and not in groups). Outside of physiotherapy times participants are encouraged to rest in the day hospital and complete a workbook. A single independent physiotherapist will be trained to deliver the intervention.

The participant (+/- family member) will attend an initial meeting with the consultant neurologist and the treating physiotherapist. The neurologist will perform a brief neurological assessment and confirm the diagnosis.

1. The diagnosis will be explained again to the patient, using the word "functional" to describe the diagnosis.
2. Physical signs of FMS will be demonstrated to the patient. This includes distractibility, Hoover's sign and entrainment.
3. The treatment programme will be explained to the patient, linking resolution of symptoms with treatment rationale.
4. The participant will attend 8-9 physiotherapy sessions over the 5 days. The intervention is a combination of education on functional motor symptoms, movement retraining and development of a self management plan.
5. After the final physiotherapy session, the participant will complete the outcome measures (Time 2) and a feedback form.

Both groups will be followed up at 6 months after recruitment to the study (Time 3). An independent assessor will administer the outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* A clinically established diagnosis of functional motor symptoms according to the Fahn-Williams criteria.
* Diagnostic investigations have come to an end.
* The patient accepts the diagnosis of functional motor symptoms.
* Symptom duration of at least six months.
* Symptoms must be sufficient to cause significant distress (subjectively described by the patient) or impairment in social, occupational or other important areas of functioning.

Exclusion Criteria:

* Unable to understand English.
* Pain, fatigue or dissociative seizures is the predominant symptom.
* Prominent untreated axis 1 disorders (e.g. anxiety or depression).
* Level of disability prevents participation in a 5 day outpatient programme (Barthel Index score less than 25/100)
* Patient unable to attend 5 consecutive days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-09; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Clinical Global Impression Scale of Change | Approximately 4 weeks after randomisation (this will be immediately after treatment for the experimental arm) and 6 months
  Self rated 5 point Likert scale of change

SECONDARY OUTCOMES:
Short Form 36 | Baseline and 6 months
Hospital Anxiety and Depression Scale | Baseline, approximately 4 weeks after randomisation and 6 months
EQ-5D-5L | Baseline, approximately 4 weeks after randomisation and 6 months
Brief Illness Perception Questionnaire | Baseline, approximately 4 weeks after randomisation and 6 months
Work and Social Adjustment Scale | Baseline, approximately 4 weeks after randomisation and 6 months
Disabilities of the Arm, Shoulder and Hand (DASH) | Baseline, approximately 4 weeks after randomisation and 6 months
  self reported questionnaire of upper limb function
Functional Mobility Scale | Baseline, approximately 4 weeks after randomisation and 6 months
  Scale of assistance required when walking 5, 50 and 500 metres.
Psychogenic Movement Disorders Rating Scale (PMDRS) | Baseline, approximately 4 weeks after randomisation and 6 months
  Blind video analysis of movement
Berg Balance Scale | Baseline, approximately 4 weeks after randomisation and 6 months
10 metre Walk Test | Baseline, approximately 4 weeks after randomisation and 6 months
  timed walk over 10 metres

OTHER OUTCOMES:
Client Services Receipt Inventory (CSRI) | Baseline and 6 month follow up
  This questionnaire collects retrospective information about the use of health and social care services, income, employment and benefits. It can be used to calculate service costs and total costs of care.

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Nielsen, Principal Investigator — UCL
Locations (1):
- The National Hospital for Neurology and Neurosurgery, London, United Kingdom

REFERENCES:
- [Derived] Nielsen G, Buszewicz M, Stevenson F, Hunter R, Holt K, Dudziec M, Ricciardi L, Marsden J, Joyce E, Edwards MJ. Randomised feasibility study of physiotherapy for patients with functional motor symptoms. J Neurol Neurosurg Psychiatry. 2017 Jun;88(6):484-490. doi: 10.1136/jnnp-2016-314408. Epub 2016 Sep 30. PMID 27694498